CLINICAL TRIAL: NCT05424055
Title: Prevention of Functional and Cognitive Impairment Through a Multicomponent Exercise Program in Hospitalized Oncogeriatric Patients
Brief Title: Prevention of Functional and Cognitive Impairment in Hospitalized Oncogeriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: ONCOGERI-ACUTE
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Hospital Acquired Condition; Debility; Aging
Keywords: Multicomponent exercise; Oncogeriatric; Hospitalization
MeSH Terms: conditions — Neoplasms; Iatrogenic Disease; Frailty

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Exercise (Experimental): The intervention will consist of a multicomponent exercise training programme, which will include supervised progressive resistance exercise training, balance training, and walking for 3 consecutive days. During the training period, patients will be trained in 20-minute sessions twice a day (morning and evening).
  Interventions: Behavioral: Multicomponent exercise
- Usual care (No Intervention): Participants randomly assigned to the usual care group will receive normal hospital care, including physical rehabilitation when needed

INTERVENTIONS:
Behavioral: Multicomponent exercise — The intervention will consist of a multicomponent exercise training programme, which will include supervised progressive resistance exercise training, balance-training and walking for 3 consecutive days. During the training period, patients will be trained in 20-minute sessions twice a day (morning and evening). The supervised multicomponent exercise training programme will be comprised of upper and lower body strengthening exercises, tailored to the individual's functional capacity, using weight machines and aiming for 2-3 sets of 8-10 repetitions at an intensity of 40-60 % of 1RM (Matrix, Johnson Health Tech, Ibérica, S.L., Madrid, Spain) combined with balance and gait retraining exercises that will progress in difficulty and functional exercises, such as rises from a chair. The second part of the session will consist of functional exercises such as knee extension and flexion, hip abduction, balance movements, and daily walking in the hospital.
  Arms: Multicomponent Exercise

SUMMARY:
Hospitalized older patients usually remain bedridden for many hours and this may lead to the appearance of unwanted negative consequences, such as cognitive or physical decline upon discharge. Our study will analyze whether an intervention consisting of a multicomponent training programme applied to patients over the age of 60 who are hospitalized for acute medical conditions in an Oncology Department of a tertiary hospital improves functional capacity and cognitive function. A total of 50 hospitalized older adult patients will be recruited in the Hospital Universitario de Navarra, Pamplona, Spain. The participants will be randomized and included in an exercise intervention (n = 25) or a control (n = 25) group (hospital usual-care). The intervention consists of a multicomponent exercise training programme that will take place for 3 consecutive days (2 sessions/day). The control group will receive usual hospital care, which will include physical rehabilitation when needed. Functional and cognitive impairment after and during acute hospitalization in older adults are major determinants of the later need for health resources. If our hypothesis is correct and shows that a multicomponent, individualized and progressive exercise programme is an effective therapy for improving the functional capacity of acutely hospitalized older patients compared to usual care, a change in the current system of hospitalization may be justified in oncogeriatric patients with medical conditions

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Barthel Index ≥60 points
* Able to ambulate (with/without assistance)
* Sign the informed consent
* Able to communicate

Exclusion Criteria:

* Expected length of stay < 6 days
* Terminal illness
* Very severe cognitive decline (i.e., GDS 7)
* Uncontrolled arrhythmias, acute pulmonary embolism, acute myocardial infarction or limb bone fracture in the past 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Change in functional capacity: Short Physical Performance Battery test (SPPB; Spanish versión) | 12 months
  The change in SPPB measured at baseline and follow-up (a measure of balance, gait, and rising from a chair) Minimum 1 Maximum 12 Higher scores mean a better outcome
Change in cognitive function: Minimental State Evaluation (MMSE; Spanish version) | 12 months
  The change in MMSE will be measured at baseline and follow-up. Minimum 1 Maximum 35 Higher scores mean a better outcome

SECONDARY OUTCOMES:
Change in functional capacity: Barthel Index (spanish version) | 12 months
  The change in Barthel Index measured at baseline and follow-up (a measure of Basic Activities of Daily Living) Minimum 0 Maximum 100 Higher scores mean a better outcome
Changes in handgrip strength (dominant hand) | 12 months
  The change in handgrip strength at baseline and follow-up
Gait ability will be assessed using the 6-metre gait velocity test (GVT) | 12 months
  The change in gait velocity test measured at baseline and follow-up
Changes in mood status: the 15-item Yesavage Geriatric Depression Scale (GDS-VE), Spanish version | 12 months
  The change in Yesavage Geriatric Depression Scale measured at baseline and follow-up
Changes in the Trail Making Test (TMT) part A | 12 months
  The change in Trail Making Test measured at baseline and follow-up. Minimum 0 Results are reported as the number of seconds required to complete the task; higher scores reveal greater impairment.
Dual task GVT (verbal GVT and arithmetic GVT) | 12 months
  The change in Dual task measured at baseline and follow-up. During the verbal dual-task test the investigarors will measure the gait velocity while participants name animals aloud. The cognitive score wil be measured by counting the number of animals named (verbal dual task) or by counting the numbers that were stated (arithmetic dual task) and the errors in each task. Minimum 0 Higher scores reveal greater impairment.
Changes in the quality of life measured by the Spanish version of the EuroQol-5 Dimension (EQ-5D) questionnaire | 12 months
  The change in EuroQol-5 Dimension (EQ-5D) questionnaire, measured at baseline and follow-up.
  The EQ records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine' Minimum 0 Maximum 100 Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: NICOLA MARTINEZ-VELILLA, PhD, Principal Investigator — Hospital of Navarra
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available upon reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of the first article. No limit of time for reasonable requests